CLINICAL TRIAL: NCT02031744
Title: A Randomized, Phase III, Multicenter, Double-Blind, Placebo-Controlled Study Evaluating the Efficacy and Safety of Onartuzumab (MetMAb) in Combination With Erlotinib as Second- or Third-Line Treatment for Patients With MET-Positive Incurable Stage IIIB/IV Non-Small Cell Lung Cancer
Brief Title: A Study of the Efficacy and Safety of MetMAb Combined With Tarceva in Patients With Met-Positive Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YO28345
Record Dates: First submitted 2014-01-08; First posted 2014-01-09 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; onartuzumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- erlotinib [Tarceva] + placebo (Placebo Comparator)
  Interventions: Drug: erlotinib [Tarceva]; Drug: Placebo
- erlotinib [Tarceva] + onartuzumab [MetMAb] (Experimental)
  Interventions: Drug: erlotinib [Tarceva]; Drug: Onartuzumab [MetMAb]

INTERVENTIONS:
Drug: erlotinib [Tarceva] — 150 mg oral administration once daily
Drug: Placebo — 15 mg/kg intravenous administration every 3 weeks
  Arms: erlotinib [Tarceva] + placebo
Drug: Onartuzumab [MetMAb] — 15 mg/kg intravenous administration every 3 weeks
  Arms: erlotinib [Tarceva] + onartuzumab [MetMAb]

SUMMARY:
This randomized, Phase III, double-blind, placebo-controlled study will evaluate the safety and efficacy of MetMAb (onartuzumab) in combination with Tarceva (erlotinib) compared with treatment with Tarceva alone in patients with incurable Met-positive non-small cell lung cancer (NSCLC). Patients will be randomized in a 2:1 ratio to receive either MetMAb + Tarceva or placebo + Tarceva. Tarceva (150 mg) will be given orally once daily, and MetMAb (15 mg/kg) will be given intravenously every 3 weeks. Treatment will continue until disease progression, unacceptable toxicity, a decision to discontinue, or death occurs. Total study length is expected to be around 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years or older.
* Patients with an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Histologically confirmed incurable Stage IIIB/IV NSCLC tumor.
* Met-positive status and results of epidermal growth factor receptor (EGFR)-activating mutation testing.
* Available tumor tissue sample or agreement to take such a sample.
* Radiographic evidence of disease. Lesions must be outside a previous radiotherapy field if they are the sole site of disease, unless disease progression has occurred at that site since radiation.
* Prior treatment with at least one platinum-based line of treatment for locally advanced, unresectable/inoperable disease or metastatic disease, and no more than one additional line of chemotherapy treatment, defined as follows:
* Adjuvant/neoadjuvant chemotherapy or chemoradiation counts as a line of therapy if < 12 months have elapsed between the last dose and the date of recurrence. Combined treatment with chemotherapy and radiation constitutes a single regimen; surgery is not considered a regimen.
* Cytotoxic maintenance therapy that differs from first-line therapy is considered an additional line of therapy. However, changes in treatment due to intolerance or excessive toxicity are not considered an additional regimen.
* The last dose of prior chemotherapy must have been given >/= 21 days prior to Day 1 (>/= 14 days for vinorelbine or other vinca alkaloids or gemcitabine).
* Anti-cancer agents used for pleurodesis are not counted as a line of therapy.
* Prior radiation therapy is allowed provided the patient has recovered from any toxic effects and >/= 7 days have elapsed between the last session and randomization.
* Patients must use effective contraception throughout the trial and until 3 months after the last dose.

Exclusion Criteria:

* More than 30 days expsoure to an EGFR inhibitor or a known EGFR-toxicity resulting in dose modifications.
* Prior exposure to agents targeting either the HGF or MET pathway, including but not limited to crizotinib, cabozantinib, ficlatuzumab, rilotumumab, and tivantinib.
* Pleural effusion, pericardial fluid, or ascites requiring drainage every other week or more frequently.
* Brain metastases or spinal cord compression that were not definitively treated with surgery and/or radiation or that were previously diagnosed and treated without evidence of clinically stable disease for >/= 14 days. Patients with treated central nervous system (CNS) metastases who are asymptomatic and on a stable dose of corticosteroid for >/= 14 days prior to randomization are eligible.
* History of another cancer in the previous 5 years, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin cancer, stage I uterine cancer, or other cancers that are curable.
* Life expectancy < 12 weeks.
* Radiographically visible interstitial lung disease (ILD) or a history of it. History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
* Inadequate hematologic, biological, or organ function.
* Significant history of cardiac disease.
* Serious active infection at the time of randomization or other serious underlying medical conditions that would impair the ability of the patient to receive protocol treatment, including positive HIV or active hepatitis B or C infections, significant gastrointestinal abnormalities, uncontrolled diabetes.
* Any inflammatory changes to the surface of the eye.
* Inability to take oral medication, need for intravenous alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease.
* Pregnant or breast-feeding women.
* Any major surgery within 2 weeks prior to randomization.
* Inability to understand the language(s) in which the HRQOL questionnaires are available.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 530 (Estimated)
Dates: Start 2014-01-22 (Actual); Primary Completion 2016-01-06 (Actual); Study Completion 2016-01-06 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | Up to 36 months
Incidence of adverse events | Up to 33 months

SECONDARY OUTCOMES:
Progression-free survival (PFS), defined as time from randomization until progression as measured by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 or death. | Up to 36 months
Overall response rate (ORR), as measured by RECIST v1.1 | Up to 36 months
Health-related quality of life (HRQOL) as measured by the European Organization for the Research and Treatment of Cancer (EORTC) assessments | Up to 33 months
Incidence of anti-therapeutic antibodies against MetMAB | Up to 33 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (8):
- China (8):
  - The Affiliated Hospital of Military Medical Sciences(The 307th Hospital of Chinese PLA), Beijing
  - Jilin Cancer Hospital, Changchun
  - Southwest Hospital , Third Military Medical University, Chongqing
  - Third Affiliated Hospital of Third Military Medical University, Chongqing
  - Sun Yet-sen University Cancer Center, Guangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Jiangsu Cancer Hospital, Nanjing